CLINICAL TRIAL: NCT03604978
Title: A Phase I/II Study of Nivolumab Plus or Minus Ipilimumab in Combination With Multi-Fraction Stereotactic Radiosurgery for Recurrent High-Grade Radiation-Relapsed Meningioma
Brief Title: Nivolumab and Multi-fraction Stereotactic Radiosurgery With or Without Ipilimumab in Treating Patients With Recurrent Grade II-III Meningioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01560; NCI-2018-01560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 201901009; 10186 (Other: Yale University Cancer Center LAO); 10186 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-07-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Grade 2 Meningioma; Grade 3 Meningioma; Recurrent Meningioma
MeSH Terms: conditions — Meningioma | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (nivolumab, radiosurgery) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo multi-fraction stereotactic radiosurgery on days 1, 3, and 5. Patients undergo brain MRI and blood sample collection throughout the study. Patients may also undergo ECHO as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Radiation: Stereotactic Radiosurgery
- Cohort B (nivolumab, ipilimumab, radiosurgery) (Experimental): Patients receive nivolumab IV over 30 minutes every 2 weeks for 12 doses (6 months) and then every 4 weeks for additional 6 months. Patients also receive ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 6 weeks for 4 doses in the absence of disease progression or unacceptable toxicity. Patients undergo multi-fraction stereotactic radiosurgery on days 1, 3, and 5. Patients undergo brain MRI and blood sample collection throughout the study. Patients may also undergo ECHO as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Cohort B (nivolumab, ipilimumab, radiosurgery)
Procedure: Magnetic Resonance Imaging — Undergo brain MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Radiation: Stereotactic Radiosurgery — Undergo multi-fraction stereotactic radiosurgery
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This phase I/II trial studies the side effects and best dose of nivolumab when given together with multi-fraction stereotactic radiosurgery and to see how well they work with or without ipilimumab in treating patients with grade II-III meningioma that has come back (recurrent). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. Giving nivolumab and multi-fraction stereotactic radiosurgery with or without ipilimumab may work better in treating patients with grade II-III meningioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the maximum tolerated combination and safety profile of multi-fraction radiosurgery with concurrent nivolumab plus or minus ipilimumab for recurrent radiation-relapsed high-grade meningioma. (Phase I) II. To evaluate the objective response rate (ORR), either complete response or partial response as assessed on magnetic resonance imaging (MRI) per the modified Macdonald Criteria, of multi-fraction radiosurgery with concurrent nivolumab plus or minus ipilimumab for recurrent radiation-relapsed high-grade meningioma. (Phase II)

SECONDARY OBJECTIVE:

I. To evaluate duration of overall response, progression-free survival (PFS) and overall survival (OS) of recurrent radiation-relapsed high-grade meningioma patients treated with the combination of multi-fraction radiosurgery and nivolumab plus or minus ipilimumab.

CORRELATIVE OBJECTIVES:

I. To analyze the immunophenotype changes of peripheral T-cells during the treatment with multi-fraction radiosurgery in combination with nivolumab plus or minus ipilimumab.

II. To perform molecular profiling assays on pretreatment/baseline archival tumor, including, but not limited to, whole exome sequencing (WES) and messenger ribonucleic acid (RNA) sequencing (RNAseq), in order to IIa. Identify potential predictive and prognostic biomarkers (such as neoantigen signature or mutation burden) beyond any genomic alteration by which treatment may be assigned.

IIb. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

III. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

IV. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the National Cancer Institute Early-Phase and Experimental Clinical Trials Biospecimen Bank (EET Biobank).

OUTLINE: This is a phase I, dose-escalation study of nivolumab followed by a phase II study. Patients are randomized to 1 of 2 cohorts.

COHORT A: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo multi-fraction stereotactic radiosurgery on days 1, 3, and 5.

COHORT B: Patients receive nivolumab IV over 30 minutes every 2 weeks for 12 doses (6 months) and then every 4 weeks for additional 6 months. Patients also receive ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 6 weeks for 4 doses in the absence of disease progression or unacceptable toxicity. Patients undergo multi-fraction stereotactic radiosurgery on days 1, 3, and 5.

Patients undergo brain MRI and blood sample collection throughout the study. Patients may also undergo echocardiography (ECHO) as clinically indicated.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed World Health Organization (WHO) grade II-III meningioma which has relapsed after prior radiation therapy with radiologically progressive or recurrent disease
* Patients must have measurable disease, defined as at least 1 lesion that can be accurately measured in at least one dimension as >= 1 cm on brain magnetic resonance imaging (MRI) but with the maximum dimension =< 5 cm OR gross tumor volume < 20 cm^3. All the relapsed disease would need to be eligible to be treated with reirradiation
* Patients must have at least one prior surgery with available archival formalin-fixed paraffin-embedded (FFPE) tumor blocks of the initial or recurrent meningioma. If there are multiple tumor blocks from multiple surgeries, the most recent tumor block (and ideally of the relapsed tumor after initial radiation therapy) should be submitted. If a tumor block is not available, an alternative of 20-30 unstained slides may be submitted instead. Annotation regarding whether the tumor block is before or after initial radiation therapy should be provided
* Prior initial radiation therapy may include external beam radiation or radiosurgery, or combination of both. However, the total dose of prior radiation exposure to the site of recurrent tumor (for consideration of re-irradiation) cannot be more than 70 Gy. The duration since the previous radiation exposure to the site of reirradiation need to be at least 6 months
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 x institutional normal
* The effects of nivolumab and/or ipilimumab on the developing human fetus are unknown. For this reason and because radiation therapy is known to be teratogenic, women of childbearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of investigational drug. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
  * WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 100 days
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document or, if decision-making capacity is impaired, consent of a legally authorized representative (e.g., spouse, adult child, live-in caretaker).

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have had radiation therapy (to the site of reirradiation) within 6 months prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1); however, alopecia, sensory neuropathy =< grade 2, or other =< grade 2 not constituting a safety risk based on the investigator's judgment are acceptable
* Patients who are receiving any other investigational agents
* Patients who have previous treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab and/or ipilimumab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Current use of immunosuppressive medication (EXCEPT for the following: Intranasal, inhaled, topical steroids, or local steroid injection [e.g. intra-articular injection]; systemic corticosteroids at doses =< 4 mg/day of dexamethasone or equivalent; steroids as premedication for hypersensitivity reactions [e.g. computed tomography (CT) scan premedication])
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. However, patients with human immunodeficiency virus (HIV) on stable therapy with minimal viral loads and patients with hepatitis B and hepatitis C who have received treatment with minimal viral loads will be eligible
* Pregnant women are excluded from this study because radiation therapy is teratogenic and that the effects of nivolumab and/or ipilimumab on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and/or ipilimumab, breastfeeding should be discontinued if the mother is treated with nivolumab and/or ipilimumab
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

  * Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Prior organ transplantation including allogeneic stem cell transplantation
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Live vaccination within 4 weeks of the first dose of nivolumab and while on trial is prohibited except for administration of inactivated vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated combination of radiosurgery and nivolumab plus or minus ipilimumab (Phase I) | Up to 100 days
Incidence of adverse event profile (Phase I) | Up to 100 days
  Will be evaluated by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The number and percentage of subjects experiencing each type of adverse event will be tabulated by severity, and relationship to treatment. If appropriate, confidence intervals will be used to characterize the precision of the estimate. A complete listing of adverse events will also be tabulated, and will provide details including severity, relationship to treatment, onset, duration, and outcome. Laboratory data measured on a continuous scale will be characterized by summary statistics (mean and standard deviation).
Objective response rate (Phase II) | From the start of treatment through at least two years of follow-up
Objective radiological response (Phase II) | Up to 100 days
  Will include either complete response or partial response as assessed on magnetic resonance imaging per the modified Macdonald Criteria. 80% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Progression-free survival | From the start of treatment to 6 months and 2 years
  80% confidence intervals will be assessed using Kaplan-Meier product limit methods.
Overall survival | From the start of treatment through at least two years of follow-up
  80% confidence intervals will be assessed using Kaplan-Meier product limit methods.
Duration of overall response | From the start of treatment through at least two years of follow-up

OTHER OUTCOMES:
Deoxyribonucleic acid sequencing | Up to 100 days
  Will be explored by comparing the differences in theses biomarkers between responders versus non-responders using t-test or Mann-Whitney rank-sum test as appropriate. Permutation test will be used to determine whether the observed difference is larger than might be expected by chance, while the null distribution of test statistics will be generated using 10,000 permutation samples where the response status will be randomly re-shuffled. The observed test statistics will be compared to the null distributions. For each outcome, the permuted p-value will be the fraction of permuted samples that resulted in a small statistic than the original sample.
Ribonucleic acid expression | Up to 100 days
  Will be explored by comparing the differences in theses biomarkers between responders versus non-responders using t-test or Mann-Whitney rank-sum test as appropriate. Permutation test will be used to determine whether the observed difference is larger than might be expected by chance, while the null distribution of test statistics will be generated using 10,000 permutation samples where the response status will be randomly re-shuffled. The observed test statistics will be compared to the null distributions. For each outcome, the permuted p-value will be the fraction of permuted samples that resulted in a small statistic than the original sample.
Neoantigen signature | Up to 100 days
  Will be explored by comparing the differences in theses biomarkers between responders versus non-responders using t-test or Mann-Whitney rank-sum test as appropriate. Permutation test will be used to determine whether the observed difference is larger than might be expected by chance, while the null distribution of test statistics will be generated using 10,000 permutation samples where the response status will be randomly re-shuffled. The observed test statistics will be compared to the null distributions. For each outcome, the permuted p-value will be the fraction of permuted samples that resulted in a small statistic than the original sample.
Changes of peripheral T-cells | Baseline up to 100 days
  Each T-cell subset will be quantified as a percentage of the overall T-cell population by normalizing to CD3+ cells. Linear mixed model for repeated measurement data will be used to assess the change over time as well as the differences between subgroups (e.g., responders vs. non-responders) for immunogenicity and other biomarkers (i.e., frequency of CD8+Ki67+PD1+ T-cells, etc.). Receiver operating characteristic (ROC) curves will also be used to assess the overall predictive ability and to explore the optimal cut-off points for baseline biomarkers to differentiate responders versus non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, Principal Investigator — Yale University Cancer Center LAO
Locations (29):
- United States (29):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm